CLINICAL TRIAL: NCT03919526
Title: The Safety and Clinical Efficacy of Human CD19/CD22 Bispecific Chimeric Antigen Receptor (CAR)-T Cell Therapy for Subjects With Measurable Residual Disease(MRD)-Positive B Cell Acute Lymphoblastic Leukemia
Brief Title: Anti-CD19/CD22 Bispecific Chimeric Antigen Receptor（CAR)-T Cell Therapy for Measurable Residual Disease(MRD) Positive ALL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, principal investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-CAR-T MRD+ALL
Record Dates: First submitted 2019-04-07; First posted 2019-04-18 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: MRD-positive; Acute Lymphoblastic Leukemia
Keywords: CD19/CD22; Bispecific CAR-T; leukemia; MRD-positive; B-ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/CD22 CAR-T cells (Experimental): Administration with anti-CD19/ CD22 CAR-T cells in the MRD-positive ALL patients.
  Interventions: Biological: anti-CD19/CD22 CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-CD19/CD22 CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-CD19 and anti-CD22 CARs
Drug: Fludarabine — 30mg/m2/d
Drug: Cyclophosphamide — 300mg/m2/d

SUMMARY:
To evaluate the safety and efficacy of CD19/CD22 Bispecific chimeric antigen receptor (CAR)-T for the treatment of measurable residual disaese (MRD)-positive B cell acute lymphoblastic leukemia. Patients will be given a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of CD19/CD22 CAR+ T cells.

DETAILED DESCRIPTION:
Participants with MRD-positive B cell acute lymphoblastic leukemia can participate if all eligibility criteria are met. Tests required to determine eligibility include disease assessments, a physical exam, Electrocardiograph, CT/MRI , and blood draws. Participants receive chemotherapy prior to the infusion of CD19/CD22 CAR+ T cells. After the infusion, participants will be followed for side effects and effect of CD19/CD22 CAR+ T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* (1) CD19 positive/CD22 positive, or CD19-CD22 positive B-cell acute lymphoblastic leukemia;
* (2)18 to 70 Years Old, Male and female;
* (3) Expected survival > 12 weeks;
* (4) ECOG score 0-2;
* (5) Bone marrow examination clearly diagnosed as B-cell acute lymphoblastic leukemia and who met one of the following conditions:

  1. Recurrent patients who achieves MRD-positive CR or CRi after standard therapy;
  2. Those who achieves CR, but failed to achieve MRD-negative after at least 2 courses of consolidation therapy;
  3. For Ph-positive ALL patients, a history of at least one TKI application is required in addition to two standard chemotherapy treatments
* (6) The venous access required for collection can be established and mononuclear cell collection can be determined by the investigators;
* (7) Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Creatinine is in the normal range;
  2. Left ventricular ejection fraction >50%;
  3. Baseline oxygen saturation>92%;
  4. Total bilirubin ≤ 2×ULN;
  5. ALT and AST ≤ 2.5×ULN;
* (8) Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

* (1) Malignant tumors other than acute lymphoblastic leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection;
* (2) Subjects with positive HBsAg or HBcAb and peripheral blood HBV DNA titer detection ≥ 1 × 102 copy number / L; HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; CMV DNA positive; syphilis positive;
* (3) Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
* (4) Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
* (5) Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* (6) Received CAR-T treatment or other gene therapies before enrollment;
* (7) Patients with symptoms of central nervous system;
* (8) Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell transfusion;
* (9) The investigators consider other conditions unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Safety measured by occurence of study related adverse effects defined by NCI CTCAE5.0 | 28 days post infusion
  Safety measured by occurence of study related adverse effects defined by NCI CTCAE5.0

SECONDARY OUTCOMES:
MRD clearance | 3 months post infusion
  MRD clearance
Content of CD19 positive B-cells in peripheral blood | 3 months post infusion
  Content of CD19 positive B-cells in peripheral blood
Content of CAR-T related cytokines positive T cells in circulation | 3 months post infusion
  Content of CAR-T related cytokines positive T cells in circulation
Total response rate (ORR) after administration | 3 months post infusion
  Total response rate (ORR) after administration including complete response(CR) and partial response(PR)
Duration of remission (DOR) after administration | 2 years post infusion
  Duration of remission (DOR) after administration
Overall Survival (OS)after administration | 2 years post infusion
  Overall Survival (OS)after administration

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No